CLINICAL TRIAL: NCT01557075
Title: Effects of High-dose Statin Treatments on Patients With Aspirin Mono Antiplatelet Therapy 12-months After Drug-eluting Stents Implantation: a Randomized Controlled Study
Brief Title: Aspirin Mono Therapy 12-months After Drug-eluting Stents Implantation
Acronym: statin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Myeong-Ki Hong, Professor of cardiology, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2010-0298
Record Dates: First submitted 2012-03-12; First posted 2012-03-19 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Drug-eluting Stent (DES)
Keywords: High dose statin
MeSH Terms: interventions — Atorvastatin; Pravastatin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin group (Active Comparator): Atorvastatin 40 mg daily for 12 months after randomization
  Interventions: Drug: Atorvastatin (High dose statin treatment)
- Pravastatin group (Active Comparator): Pravastatin 20mg daily for 12 months after randomization
  Interventions: Drug: Pravastatin (High dose statin treatment)

INTERVENTIONS:
Drug: Atorvastatin (High dose statin treatment) — Patients will be randomly assigned to the type of statins. Randomization of statin therapy will be done 1:1 to one of two different statins on the web-based program
  * Atorvastatin 40 mg daily for 12 months after randomization
  Other Names: DES-statin
  Arms: Atorvastatin group
Drug: Pravastatin (High dose statin treatment) — Patients will be randomly assigned to the type of statins. Randomization of statin therapy will be done 1:1 to one of two different statins on the web-based program
  Pravastatin 20mg daily for 12 months after randomization
  Arms: Pravastatin group

SUMMARY:
The purpose of this study is to determine whether high dose statin therapy in patients with aspirin mono antiplatelet therapy who had received drug-eluting stent (DES) previously and were free of the adverse cardiac events during the first 12 months could be superior over pravastatin therapy in the prevention of late adverse cardiac and cerebrovascular events during the additional 12 months.

Study Design.

DETAILED DESCRIPTION:
Objective: To determine whether high dose statin therapy in patients with aspirin mono antiplatelet therapy who had received drug-eluting stent (DES) previously and were free of the adverse cardiac events during the first 12 months could be superior over pravastatin therapy in the prevention of late adverse cardiac and cerebrovascular events during the additional 12 months.

Study Design

* Prospective, randomized, multi-center study of each 1000 subjects enrolled.
* Eligible subjects will be randomized 1:1 to a) atorvastatin 40 mg (n=1000) vs. b) pravastatin 20 mg/day (n=1000). All subjects will be followed for 1 year after randomization. Additional long-term follow-up (2- or 3-year) will be preceded in the next plan after 1-year study period.
* Subjects with coronary artery diseases who meet all inclusion and exclusion criteria will be included Clinical and laboratory follow-up should be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had previously received DES at least 12 months(±2month) ago
2. Patients who were free of death, MI, stroke, repeat revascularization, or ST within first 12 months after DES implantation
3. Patients with mono antiplatelet therapy with only aspirin after
4. Age 20 years of older
5. Patients with signed informed consent

Exclusion Criteria:

1. History of DES or BMS implantation within 10 months
2. Patients who required the continuing dual antiplatelet therapy or additional other types of antithrombotics or antiplatelets such as cilostazol or ticlopidine, etc besides aspirin after DES implantation
3. Patients who could not be prescribed aspirin or statins due to contraindication or severe side effects
4. Pregnant women or women with potential childbearing
5. Life expectancy ≤ 2 year

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2010-07; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
the composite of death from any cause | 12 months after randomization
  Occurrence of the composite of death from any cause, MI, target vessel revascularization (TVR, either by PCI or CABG), non-TVR, stent thrombosis (ST), peripheral artery intervention, deterioration of renal function, stroke or admission for significant clinical cardiac events for 12 months following the randomization to the assigned statin therapy.

SECONDARY OUTCOMES:
cardiac or non-cardiac death | 12month
  1. Major determinant for the occurrence of major events(death,MI,TVR,ST)
  2. Comparisons of the occurrence of major events according to the attainment of recommended LDL-C goal on current lipid guideline
  3. Association between laboratory test and clinical outcomes;
  4. Sub-study according to the subsets of disease
  5. Association between parameters at index procedure and clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Myeong-Ki Hong, MD.PhD., Principal Investigator — Severance Hospital
Locations (1):
- Hong Myeong-Ki, Seoul, South Korea

REFERENCES:
- [Derived] Im E, Cho YH, Suh Y, Cho DK, Her AY, Kim YH, Lee K, Kang WC, Yun KH, Yoo SY, Cheong SS, Shin DH, Ahn CM, Kim JS, Kim BK, Ko YG, Choi D, Jang Y, Hong MK. High-intensity Statin Treatments in Clinically Stable Patients on Aspirin Monotherapy 12 Months After Drug-eluting Stent Implantation: A Randomized Study. Rev Esp Cardiol (Engl Ed). 2018 Jun;71(6):423-431. doi: 10.1016/j.rec.2017.06.008. Epub 2017 Jul 14. English, Spanish. PMID 28716428